CLINICAL TRIAL: NCT03026725
Title: Effect of Tri Calcium Phosphate Paste on Efficacy and Postoperative Sensitivity Associated With At-Home Vital Tooth Whitening Using 20% Carbamide Peroxide 'A Randomized Controlled Study'
Brief Title: Effect of Tri Calcium Phosphate on Efficacy and Sensitivity With Vital Tooth Whitening Using 20% Carbamide Peroxide
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UDDS-OperDent-03-2016
Record Dates: First submitted 2017-01-18; First posted 2017-01-20 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Tooth Sensitivity
Keywords: tooth sensitivity; tri calcium phosphate; at-home whitening
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tri-calcium Phosphate (Experimental): clinpro tooth creme, i.e. Tri-calcium Phosphate, for 30 min/day after bleaching 4h with carbamide peroxide 20%
  Interventions: Other: Tri-calcium Phosphate
- Placebo (Placebo Comparator): a placebo creme will be applied for 30 min/day after bleaching 4h with carbamide peroxide 20%
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Tri-calcium Phosphate — A paste contains Tri Calcium Phosphate & Fluoride
  Other Names: ( Clinpro™ Tooth Crème, 3M ESPE, USA
  Arms: Tri-calcium Phosphate
Other: Placebo — paste manufactured to mimic Clinpro, without Tri Calcium Phosphate
  Arms: Placebo

SUMMARY:
Teeth sensitivity is the most popular symptom when using At-Home tooth whitening. Tri calcium phosphate containing pastes may affect the efficacy and postoperative sensitivity associated with At-Home vital tooth whitening using 20% carbamide peroxide

DETAILED DESCRIPTION:
Subjects enrolled in this study will apply home bleaching trays with 20%carbamide peroxide 4h/day for a week, the sample will be divided into two groups : the experimental group will apply tri calcium phosphate containing paste(Clinpro) 30 min/day after bleaching treatment, the control group will apply placebo paste 30 min/day after bleaching treatment,

ELIGIBILITY:
Inclusion Criteria:

* Good dental health
* Six maxillary anterior teeth present and healthy with no restorations or carious lesions
* Teeth darker than Vita A2 shade
* No history of teeth sensitivity
* No use of a desensitizing agent or desensitizing toothpaste in the past three months

Exclusion Criteria:

* Active caries or periodontal disease
* Allergies to bleaching agent or tray material
* pregnancy and breastfeeding during the trial
* tetracycline-stained teeth or fluoride or non-vital teeth
* Smoker
* Using tooth bleaching products during the last 3 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-11; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Change in Sensitivity Status | at (1) 24 hours following application, (2) at 48 hours post-application, (3) at 72 hours post-application and (4) at seven days following application
  using a visual analog scale (VAS)

SECONDARY OUTCOMES:
Change in Color Shade | at (1) 72 hours following application , (2) one week following application, (3) two weeks following application, and (4) one month following application
  color shade change will be detected; using Vita Easy Shadeِ Advance 4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Oula Yassin, DDS, MSc,Phd, Principal Investigator — Damascus University
Locations (1):
- Damascus University, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maghaireh GA, Alzraikat H, Guidoum A. Assessment of the effect of casein phosphopeptide-amorphous calcium phosphate on postoperative sensitivity associated with in-office vital tooth whitening. Oper Dent. 2014 May-Jun;39(3):239-47. doi: 10.2341/12-527-C. Epub 2013 Oct 22. PMID 24147745
- [Background] Loguercio AD, Tay LY, Herrera DR, Bauer J, Reis A. Effectiveness of nano-calcium phosphate paste on sensitivity during and after bleaching: a randomized clinical trial. Braz Oral Res. 2015;29:1-7. doi: 10.1590/1807-3107BOR-2015.vol29.0099. Epub 2015 Aug 21. PMID 26313348
- [Background] Pintado-Palomino K, Peitl Filho O, Zanotto ED, Tirapelli C. A clinical, randomized, controlled study on the use of desensitizing agents during tooth bleaching. J Dent. 2015 Sep;43(9):1099-1105. doi: 10.1016/j.jdent.2015.07.002. Epub 2015 Jul 6. PMID 26159384
- [Background] Dawson PF, Sharif MO, Smith AB, Brunton PA. A clinical study comparing the efficacy and sensitivity of home vs combined whitening. Oper Dent. 2011 Sep-Oct;36(5):460-6. doi: 10.2341/10-159-C. Epub 2011 Aug 22. PMID 21859318
- [Background] Basting RT, Amaral FL, Franca FM, Florio FM. Clinical comparative study of the effectiveness of and tooth sensitivity to 10% and 20% carbamide peroxide home-use and 35% and 38% hydrogen peroxide in-office bleaching materials containing desensitizing agents. Oper Dent. 2012 Sep-Oct;37(5):464-73. doi: 10.2341/11-337-C. Epub 2012 May 18. PMID 22616927